CLINICAL TRIAL: NCT04866940
Title: Validation and Implementation of 3T MRI Research Protocols
Acronym: VALIDIRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: C20-28
Record Dates: First submitted 2021-04-07; First posted 2021-04-30 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequence validation (Experimental): This research aims to provide a generic framework to test the feasibility of MRI sequences requested as part of protocols, but also to optimize MRI acquisition sequences already in place, to improve image quality and reduce artifacts that can degrade the quality of images obtained.
  Interventions: Other: Sequences test

INTERVENTIONS:
Other: Sequences test — the realization of preliminary acquisitions to validate the feasibility of clinical or cognitive research protocols

SUMMARY:
The Philips 3T imager installed on the Pavillon Baudot site is an imager dedicated solely to research. It is not located in hospital premises but in INSERM premises for which an authorization for biomedical research has been granted. This equipment is part of the Technical Platform of the UMR 1214 ToNIC whose main objective is the study of the human brain and the main pathologies that affect it.

MRI is an evolving technique, which is used in many research projects. Our technical platform must follow these developments and remain at the cutting edge. One of the essential services of our technical platform is to help set up research protocols and validate acquisition sequences. This development activity is therefore located upstream of research projects involving clinical or fundamental applications. The fact that we can provide our users with a regulatory framework to carry out these development tests for their Research Involving Human Subjects project is a necessity for our research support activity.

This study aims to provide a generic framework to test the feasibility of MRI sequences requested within the framework of protocols, but also to optimize MRI acquisition sequences already in place, to improve image quality and reduce artifacts that can degrade the quality of the images obtained.

In France, there are just over 35 centers with MRI dedicated to research and therefore with a validation protocol allowing them to validate their sequences.

DETAILED DESCRIPTION:
This is a prospective monocentric research on major participants (healthy and patients). The optimization of the sequences will be carried out in an incremental way from one control to the other: for each control, several sequences will be carried out for an acquisition time not exceeding one hour of cumulated acquisition (i.e. one hour and a half including the installation and the delays between the sequences). Each sequence lasts between 5 and 20 minutes.

At the end of the examination, the images obtained will be evaluated jointly by an expert neuroradiologist and a research engineer specialized in image analysis according to the criteria mentioned above. This analysis will make it possible to determine the parameters to be modified to improve image quality and to define the acquisition parameters for the next test.

As soon as a sequence is considered optimal, it will be tested on a small number of healthy controls (≈ 5) to ensure interindividual reproducibility of image quality parameters, and then if necessary in the presence of pathology in a few patients (≈ 5).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Ability to cooperate and remain motionless for up to 1 hour (and lying down for 1.5 hours)
* Ability to understand the instructions given
* Subject who has given written and informed consent prior to any examination required by the research)
* Subject affiliated to a social security system or benefiting from an equivalent system

Exclusion Criteria:

* Persons deprived of liberty by judicial or administrative decision
* Psychiatric disorders, disorders of cognitive functions, not allowing the realization of the MRI
* Protected adults (subject to a measure of legal protection) or unable to express their consent
* Subject with Contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
in general | at the end of studies ((i.e. one hour and a half including the installation and the delays between the sequences). Each sequence lasts between 5 and 20 minutes.
  optimization of parameters acquisition in order to suppress artefact

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PAYOUX, Pr, Principal Investigator — Inserm: UMR 1214 ToNIC
Locations (1):
- UMR 1214 ToNIC INSERM, Toulouse, France

IPD SHARING:
Plan to Share IPD: No